CLINICAL TRIAL: NCT03119233
Title: The Detour Endovascular Technique for Long OcclUsive Fem-pop Revascularization - 2 Clinical Trial
Brief Title: The DETOUR 2 Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STP 203
Record Dates: First submitted 2017-04-11; First posted 2017-04-18 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single-Arm (Experimental): This is a prospective, single-arm, multi-center, international clinical investigation to evaluate the safety and effectiveness of the DETOUR System, delivery guidewires, and implant stent grafts for percutaneous femoropoliteal bypass compared to Performance Goals (PG)
  Interventions: Device: DETOUR System

INTERVENTIONS:
Device: DETOUR System — The DETOUR System is intended to improve blood flow in patients with peripheral arterial disease in symptomatic femoropopliteal lesions due to chronic total occlusions ≥ 20 cm (TASC D) that can include de novo, restenotic, or in-stent restenotic lesions; or total lesion lengths ≥24 cm that can include chronic total occlusions or a ≥70% lesion that includes de novo, restenotic or in-stent restenosis (complex TASC C).

SUMMARY:
Prospective, single-arm, multi-center, international clinical investigation to evaluate the safety and effectiveness of the PQ Bypass System to access, deliver guidewires, and implant stent grafts for a percutaneous femoropopliteal (fem-pop) bypass.

DETAILED DESCRIPTION:
The DETOUR2 study is a prospective, single-arm, multi-center, international, non-randomized, safety and effectiveness clinical investigation of the PQ Bypass system.

The PQ Bypass System is intended to improve blood flow in patients with symptomatic peripheral arterial disease due to symptomatic femoropopliteal chronic total occlusions ≥ 20 cm (TASC D) that can include de novo, restenotic, or in-stent restenotic lesions; or Symptomatic femoropopliteal lesions ≥ 24 cm (total lesion length) that can include a chronic total occlusion or a ≥70% lesion that includes de novo, restenotic or in-stent restenosis (complex TASC C), with reference vessel diameters ranging from 5.0 - 6.7 mm, by investigator visual assessment.

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to meet the following inclusion criteria in order to be considered eligible for participation in the study:

General Inclusion Criteria

1. Age > 18 and ≤ 90 years of age.
2. Willing and able to provide informed consent.
3. Subject is willing to undergo all follow-up assessments according to the specified schedule over 36 months.

   Clinical Inclusion Criteria
4. Chronic, symptomatic lower limb ischemia defined as Rutherford clinical categories 3, 4, or 5.
5. Venous Clinical Severity Score < 3.
6. Subject is a suitable candidate for angiography and endovascular intervention and, if required, is eligible for standard surgical repair.

   Angiographic Inclusion Criteria
7. Symptomatic femoropopliteal chronic total occlusions ≥ 20 cm (TASC D) that can include de novo, restenotic, or in-stent restenotic lesions; or Symptomatic femoropopliteal lesions ≥ 24 cm (total lesion length) that can include a chronic total occlusion or a ≥70% lesion that includes de novo, restenotic or in-stent restenosis (complex TASC C), by investigator visual assessment.
8. Reference vessel diameter ≥ 4.5 and ≤ 6.7 mm, by investigator visual assessment.
9. Subject has a patent popliteal artery (<50% stenosis) distal to the landing zone
10. Able to successfully access the SFA origin for entry of the crossing device.
11. At least one patent infrapopliteal vessel (<50% stenosis) with run-off to the ankle or foot.
12. A significant stenosis (≥ 50%) or occlusion of an ipsilateral, inflow artery (e.g. aortoiliac, common femoral) must be successfully treated (use of investigational treatment prohibited) prior to treatment of the target lesion. Successful treatment is defined as no complications and less than 30% residual stenosis following intervention.

General Exclusion Criteria

1. Participating in another investigational clinical study.
2. Anticipated life expectancy less than 1 year or medical comorbid condition(s) that could limit the subject's ability to comply with the requirements of the trial.
3. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.

   Clinical Exclusion Criteria
4. History of deep vein thrombosis on either limb.
5. Thrombophlebitis, within the previous 30 days.
6. 6. Planned major amputation of the target limb, including minor amputation (above the ankle).
7. Prior distal amputation (above the transmetatarsal) of the target limb.
8. Known or suspected active infection at the time of the procedure (e.g., WIfI foot infection grade 3: Severe infection. Local infection with systemic inflammatory response syndrome [SIRS])
9. Rutherford clinical category 0, 1, 2 or 6.
10. Has acute or chronic renal disease with GFR ≤ 30 ml/min per 1.73 m2 and/or elevated serum creatinine >2.5mg/dL (220µmol/L) or on dialysis.
11. Known hypersensitivity/allergy to the investigational devices and/or required pharmacotherapy that cannot be safely managed.
12. Morbid obesity that does not allow for safe vascular access or imaging.
13. Subject has a known coagulopathy or has bleeding diatheses, thrombocytopenia with platelet count less than 100,000/microliter or INR > 1.8.
14. Requires coronary or peripheral procedure within 30 days prior to or planned within 30 days post treatment of the target lesion.
15. Has a known history of intracranial bleeding or aneurysm, myocardial infarction or stroke within the last 3 months.
16. Subject is pregnant or breast-feeding. Angiographic Exclusion Criteria
17. Stent within 3 cm of SFA ostium.
18. Previous bypass surgery on the target limb.
19. Subject has significant disease or obstruction (≥50%) of the inflow tract that has not been successfully treated at the time of the index procedure (success measured as ≤30% residual stenosis, without complication)
20. Presence of aneurysm or acute thrombus in the target limb.
21. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2023-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Mustapha, MD, Principal Investigator — Advanced Cardiac and Vascular Amputation Prevention Centers; Sean Lyden, MD, Principal Investigator — The Cleveland Clinic
Locations (34):
- United States (30):
  - HonorHealth, Scottsdale, Arizona
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Bay Area Vein and Vascular, Burlingame, California
  - Community Hospital of the Monterrey Peninsula, Monterey, California
  - Advanced Cardiovascular Specialists, Mountain View, California
  - Denver VA Medical Center, Denver, Colorado
  - The Vascular Experts, Darien, Connecticut
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Baptist Hospital Miami, Miami, Florida
  - Christie Clinic, Champaign, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - McLaren Bay Region Hospital, Bay City, Michigan
  - Advanced Cardiac and Vascular Amputation Prevention Centers, Grandville, Michigan
  - Cardiac & Vascular Research Center of Nothern Michigan, Petoskey, Michigan
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - New York-Presbyterian / Columbia University Medical Center, New York, New York
  - North Caroline Hearth and Vascular- University of North Carolina Rex, Raleigh, North Carolina
  - The Christ Hospital - The Carl & Edyth Lindner Center for Research & Education, Cincinnati, Ohio
  - Cleveland Clinical Foundation, Cleveland, Ohio
  - Miriam Hospital, Providence, Rhode Island
  - Greenville Health System, Greenville, South Carolina
  - North Dallas Research Associates, Dallas, Texas
  - Texas Tech, Lubbock, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Aurora Research Institute, Milwaukee, Wisconsin
- Germany (3):
  - Klinikum Hochsauerland GmbH, Arnsberg
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Universität Leipzig, Leipzig
- Pauls Stradins Clinical University Hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment in the DETOUR 2 study was completed on 05-October-2020. All eligible subjects completed the 30-day, follow-up visit, per the protocol. Compliance at the 6, 12, and 24-month follow-up visits was 95.5%, 91.9%, and 87.05%, respectively.
Pre-assignment Details: The DETOUR 2 study enrolled subjects at 32 US and 4 OUS sites 'All Subjects' (n=202 enrolled)
Groups:
- Single Arm Intent to Treat (ITT) All Subjects: This was a single arm study, Intent to Treat (ITT) includes all subjects enrolled in the IDE Study. ITT is the primary analysis population to determine if the primary safety endpoint was met in the study.
Period: Overall Study
Arm/Group | Single Arm Intent to Treat (ITT) All Subjects
Started | 202
Completed | 202
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Intention to Treat (ITT) All Subjects: This is a prospective, single-arm, multi-center, international clinical investigation to evaluate the safety and effectiveness of the PQ Bypass System, delivery guidewires, and implant stent grafts for percutaneous femoropopliteal bypass. The primary analysis population will include 202 subjects.
Arm/Group | Single Arm Intention to Treat (ITT) All Subjects
Number analyzed (Participants) | 202
Age, Continuous [Mean (Full Range); unit: Years] | 68.9 [47 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 149
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 175
  More than one race | 2
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  Latvia | 26
  United States | 153
  Germany | 23
Rutherford clinical category [Count of Participants; unit: Participants] — Clinical scale identifying three grades of claudication and three grades of critical limb ischemia ranging from rest pain alone to minor and major tissue loss.Only subjects with Rutherford Clinical Scale Category of 3, 4 and 5, are eligible for enrollment.
  3=Severe Claudication 4=Ischemic Rest Pain 5=Minor Tissue Loss
  Participants
    Grade 3 | 157
    Grade 4 | 36
    Grade 5 | 9
Renal Insufficiency [Count of Participants; unit: Participants] — An increase in serum creatinine of ≥ 1.0 mg/dl over previous value requiring medical treatment but which does not require dialysis to resolve.
  Participants | 22
History of Smoking [Count of Participants; unit: Participants]
  Current/Previous | 184
  Never | 18
Previous Peripheral Intervention [Count of Participants; unit: Participants] | 121
History of Diabetes [Count of Participants; unit: Participants]
  Type 1 | 1
  Type 2 | 69
Congestive Heart Failure [Count of Participants; unit: Participants] | 25
Lesion Length [Mean (Standard Deviation); unit: mm] — Population: Lesion Length (Normal to Normal, mm) continuous variables presented as mean ± SD (N) where N is the number of subjects with available data.
  mm
    number analyzed (Participants) | 196
    (all) | 327.14 (61.376)
Number of Run-Off Vessels [Count of Participants; unit: Participants] — Measure Analysis Population Description: N is the number of subjects with available data, based on CoreLab data. Population: N is the number of subjects with available data.
  Participants
    1: number analyzed (Participants) | 187
    1 | 35
    2: number analyzed (Participants) | 187
    2 | 129
    3: number analyzed (Participants) | 187
    3 | 23

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency
Description: Primary patency at 12 months as evidenced by a peak systolic velocity ratio (PSVR) ≤2.5 from DUS and no clinically-driven re-intervention within the stented segment.
Time Frame: 12 months
Population: Number at Risk/Total Number of Events
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- All Subjects Intent to Treat (ITT): Primary Patency: Kaplan Meier Estimates - All Subjects
Arm/Group | All Subjects Intent to Treat (ITT)
Number analyzed (Participants) | 135
Percentage of Participants | 72.3 [66 to 78.6]
Statistical Analysis 1: Comparison: All Subjects Intent to Treat (ITT); The primary effectiveness endpoint is defined as primary patency at 12 months as evidenced by a peak systolic velocity ratio (PSVR) ≤2.5 from DUS and no clinically-driven re-intervention within the stented segment. The primary effectiveness endpoint hypotheses are: * H0: 12-month success rate of the PQ Bypass System ≤60.4% * HA: 12-month success rate of the PQ Bypass System >60.4%; Test type: Other; Lower 97.5% Exact Confidence Limit = 68.1, 97.5% CI 1-sided [lower limit 60.9]

2. Primary Outcome: Major Adverse Events at 30 Days
Description: Freedom from a Major Adverse Event (MAE) at 30 days post-procedure (defined as any occurrence of the following events: Death, Clinically-Driven Target Lesion Revascularization (CD-TLR), Major Amputation of(above the Treated Limb,ankle), Symptomatic Deep Vein Thrombosis (DVT), Pulmonary Embolism, or procedure-related bleeding requiring any transfusion of packed red blood cells or surgery).
Time Frame: 30 days
Population: MAEs at 30 days
Measure: Number; unit: Number of Events
Groups:
- All Subjects Intent to Treat (ITT): Up to 202 subjects, excluding elective roll-ins, with atherosclerotic lesions of the native superficial femoral artery (SFA) or the superficial femoral and proximal popliteal arteries, suitable for treatment will be enrolled.
Arm/Group | All Subjects Intent to Treat (ITT)
Number analyzed (Participants) | 202
Number of Events
  MAE: number analyzed (Participants) | 185
  MAE | 14
  Death: number analyzed (Participants) | 199
  Death | 0
  CD-TLR: number analyzed (Participants) | 196
  CD-TLR | 0
  Amputation of Treated Limb: number analyzed (Participants) | 199
  Amputation of Treated Limb | 0
  Deep Vein Thrombosis (DVT): number analyzed (Participants) | 194
  Deep Vein Thrombosis (DVT) | 5
  Pulmonary Embolism (PE): number analyzed (Participants) | 199
  Pulmonary Embolism (PE) | 0
  Procedure Related Bleeding: number analyzed (Participants) | 192
  Procedure Related Bleeding | 7
Statistical Analysis 1: Comparison: All Subjects Intent to Treat (ITT); The primary safety endpoint hypotheses are: * H0: 30-day Freedom from MAE rate of the PQ Bypass System ≤84% * HA: 30-day Freedom from MAE rate of the PQ Bypass System >84%; Test type: Other — The rate of freedom from 30-day MAE is expected to be no less than 92%. Based on a PG of 84% and an estimated 30-day freedom from MAE rate of 92% for the PQ Bypass System, a sample size of 169 evaluable subjects provides 88% power to test the primary safety hypothesis at the one-sided alpha level of 0.025. The Exact Test Method and Commercial software PASS14 was used to determine the sample size; Lower 97.5% Exact Confidence Limit = 93.0, 97.5% CI 1-sided [lower limit 88.5]

3. Secondary Outcome: Stent Graft Separation and Migration
Description: Stent graft separation and migration identified via ultrasound imaging
Time Frame: 30 Days
Measure: Number (95% Confidence Interval); unit: Number of Subjects
Arm/Group | All Subjects Intent to Treat (ITT)
Number analyzed (Participants) | 192
Number of Subjects
  Stent Graft Separation | 0 [0 to 1.9]
  Stent Graft Migration | 0 [0 to 1.9]
  Stent Graft Separation or Migration | 0 [0 to 1.9]

4. Secondary Outcome: Stent Graft Separation and Migration Via 12-Month X-Ray
Description: Stent graft separation and migration identified via X-ray
Time Frame: 12 Months
Population: 12 Months
Measure: Number (95% Confidence Interval); unit: Number of Subjects with available data
Arm/Group | All Subjects Intent to Treat (ITT)
Number analyzed (Participants) | 202
Number of Subjects with available data
  Stent Graft Separation: number analyzed (Participants) | 169
  Stent Graft Separation | 1 [0 to 3.3]
  Stent Graft Migration: number analyzed (Participants) | 169
  Stent Graft Migration | 3 [.4 to 5.1]
  Stent Graft Separation or Migration: number analyzed (Participants) | 169
  Stent Graft Separation or Migration | 3 [.4 to 5.1]

5. Secondary Outcome: Stent Graft Fracture Via 12-Month X-Ray
Description: Stent graft fracture identified via X-ray
Time Frame: 12-Months
Population: Based on number of subjects with available data.
Measure: Number (95% Confidence Interval); unit: Number of Subjects
Arm/Group | All Subjects Intent to Treat (ITT)
Number analyzed (Participants) | 169
Number of Subjects | 0 [0 to 2.2]

ADVERSE EVENTS:
Time Frame: All Adverse Events will be collected through 12 month follow-up. SAEs, MAEs and UADEs will be collected for the duration of the study. All device- and procedure-related events, all target limb related events, and all potential non-serious events related to study requirement medications shall be reported throughout the trial.
Description: Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related to the medical device. This includes events related to the study device or events related to the procedures involved.
Groups:
- All Subjects: All Subjects Intent to Treat (ITT)
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 14/202
Serious Adverse Events (participants affected / at risk) | 130/202
Other Adverse Events (participants affected / at risk) | 142/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=202)
Anaemia (Blood and lymphatic system disorders) | 7 (8)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Lymphoma (Blood and lymphatic system disorders) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 8 (10)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Coronary artery disease (Cardiac disorders) | 3 (3)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1)
left ventricular failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Pulmonary oedema (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Diabetes mellitus inadequate control (Endocrine disorders) | 1 (1)
Diabetic foot (Endocrine disorders) | 1 (1)
Diabetic ketoacidosis (Endocrine disorders) | 1 (1)
Hyperglycaemia (Endocrine disorders) | 1 (1)
Hypoglycaemia (Endocrine disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastroenteritis viral (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (6)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Pyloric stenosis (Gastrointestinal disorders) | 1 (1)
Stomal hernia (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (3)
Death (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 1 (1)
Organ failure (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vascular stent occlusion (General disorders) | 1 (2)
Vascular stent stenosis (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (4)
Pneumonia (Infections and infestations) | 7 (7)
Pneumonia viral (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4)
Urosepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Atheroembolism (Injury, poisoning and procedural complications) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femoral artery peforation (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Stoma complication (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site maematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Ultrasound Doppler abnormal (Investigations) | 1 (1)
Acute respiratory failure (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Humerus fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Pelvic fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper limb fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenomatous polyposis coli (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dermal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thoracic spinal stenosis (Nervous system disorders) | 1 (1)
Thrombotic stroke (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Device dislocation (Product Issues) | 2 (2)
Device malfunction (Product Issues) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Angioplasty (Surgical and medical procedures) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1)
Anaphylactic shock (Vascular disorders) | 1 (2)
Aortic aneurysm (Vascular disorders) | 1 (1)
Arterial bypass stenosis (Vascular disorders) | 2 (2)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Carotid artery stenosis (Vascular disorders) | 3 (3)
Cerebellar haemorrhage (Vascular disorders) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Compartment syndrome (Vascular disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 8 (9)
Device embolisation (Vascular disorders) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1)
Femoral artery embolism (Vascular disorders) | 1 (1)
Gastrointestinal haemorrhage (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 3 (3)
Haemorrhage intracranial (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (3)
Hypertensive emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 11 (13)
Ischaemic limb pain (Vascular disorders) | 3 (3)
Pelvic haemorrhage (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 6 (6)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
Peripheral artery haematoma (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 9 (10)
Peripheral artery restenosis (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 14 (17)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 9 (12)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
Pharyngeal haemorrhage (Vascular disorders) | 1 (1)
Retroperitoneal haematoma (Vascular disorders) | 1 (1)
Vascular stent occlusion (Vascular disorders) | 26 (31)
Vascular stent stenosis (Vascular disorders) | 11 (11)
Vascular stent thrombosis (Vascular disorders) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=202)
Anaemia (Blood and lymphatic system disorders) | 8 (9)
Atrial Fibrillation (Cardiac disorders) | 6 (6)
Oedema peripheral (General disorders) | 10 (10)
Peripheral swelling (General disorders) | 11 (11)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (20)
Deep vein thrombosis (Vascular disorders) | 27 (29)
Hypertension (Vascular disorders) | 8 (8)
Peripheral venous disease (Vascular disorders) | 6 (8)
Vascular stent occlusion (Vascular disorders) | 11 (11)
Vascular stent stenosis (Vascular disorders) | 10 (11)
Peripheral artery stenosis (Vascular disorders) | 17 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT03119233/Prot_SAP_000.pdf